CLINICAL TRIAL: NCT06659419
Title: Registry of PHAcoemulsification for Cataract Surgery
Acronym: ROPHACS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240817
Record Dates: First submitted 2024-10-16; First posted 2024-10-26 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-10

CONDITIONS: Cataract
Keywords: Cataract; Surgery; Phacoemulsification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Cataracts cause vision loss due to opacities in the lens. Cataract surgery is performed by emulsifying the nucleus of the lens. A phacoemulsifier is the machine used to deliver ultrasonic energy in the eye to fragment the lens and aspirate the debris.

In contrast to the large number of cataract procedures performed worldwide, there is surprisingly scarce data regarding the intraoperative parameters used during phacoemulsification. As new technologies are made available to surgeons, this impedes a large-scale analysis of the benefits of the advances in phacoemulsifiers. The investigators aim to establish a nationwide registry with a database of intraoperative data recorded during the cataract procedures performed with the Centurion phacoemulsifier.

The data collected would encompass all parameters recorded in the phacoemusifiers' logs, such as the energy delivered in the eye (longitudinal, torsional and other), US time, BSS volume, duration of the procedure, surgeon settings and others. The objective will be to capture data from at least 100,000 procedures/year.

DETAILED DESCRIPTION:
A nationwide registry will be established with a database of intraoperative data recorded during the cataract procedures performed with the Centurion phacoemulsifiers. The following intraoperative parameters used during the cataract surgery will be recorded and analyzed:

Primary endpoint: Ultrasound time (US time)

Exploratory endpoints:

* CDE : Cumulated dissipated Energy
* Total surgery time
* BBS volume
* Torsional and longitudinal energy
* IOP settings
* Vacuum settings Procedures performed with the Active Sentry module - where a pressure sensor is built in the phacoemulsifier handpiece will be compared to other to procedures performed without this module.

Data will be collected and analyzed from Centurions cases log extracted from at least 200 Centurions installed in France. Parameter and settings will be retrospectively analyzed.

A direct extraction of data from the machines will be processed for the analyses. No patient demographic data will be recorded.

The objective will be to capture data from at least 100,000 procedures and to run data analyses on a nationwide scale.

The database will serve as a basis to assess the technological advances aimed at reducing the amount of energy delivered in the eye, the duration of ultrasound use and overall the duration of procedures.

ELIGIBILITY:
Inclusion Criteria:

- All procedures recorded in Centurions (200 machines).

Exclusion Criteria:

* Opposition of the center to data collection.
* Complicated surgery (e.g. anterior vitrectomy) identified as such in the event log

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: No patient but procedures recorded in Centurions machine.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Description of intraoperative parameters during cataract surgery when using Active Sentry | time of the surgery
  To describe intraoperative parameters during cataract surgery when using Active Sentry compared with other handpieces in a large registry comprising at least 200 centurions (>85 benefiting from the Active Sentry upgrade). Data will be collected and analyzed from event logs extracted from 200 Centurions installed in France.
  Parameters and settings will be analyzed retrospectively.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BREZIN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Ophthalmology department - Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No